CLINICAL TRIAL: NCT03334006
Title: Prospective, Randomized Trial of Personalized Medicine With Pentaglobin® After Surgical Infectious Source Control in Patients With Peritonitis
Acronym: PEPPER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-167; 2024-513526-27-00 (EU CTIS Number); 2016-001788-34 (EudraCT Number)
Record Dates: First submitted 2017-10-27; First posted 2017-11-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Peritonitis; Sepsis; Septic Shock
Keywords: Pentaglobin®; Personalized Medicine
MeSH Terms: conditions — Peritonitis; Sepsis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: The control group receives a Standard-of-Care treatment. The intervention group is additionally treated with IgGAM (Pentaglobin®) as an add-on treatment to Standard-of-Care.
  The preparation to be provided contains (per ml solution) 50 mg human plasma proteins, of which ≥ 95 % are immunoglobulins: IgM 6 mg, IgA 6 mg and IgG 38 mg. The IgG subclass distribution is IgG1 ~ 63 %, IgG2 ~ 26 %, IgG3 ~ 4 %, IgG4 ~ 7 %.
  Pentaglobin® is administered by continuous intravenous infusion over a period of 5 day of 0.4 ml/kg body weight/hour until the total dose of 7 ml/kg body weight/day is reached.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Standard of Care treatment
- Verum arm (Active Comparator): Standard of Care treatment + Pentaglobin®
  Interventions: Drug: Pentaglobin®/Standard of Care

INTERVENTIONS:
Drug: Pentaglobin®/Standard of Care — Standard-of-Care treatment + Pentaglobin®
  Arms: Verum arm

SUMMARY:
The aim of this prospective, randomized, controlled trial is to provide evidence for adjuvant IgGAM treatment with regard to

1. Improvement of patient outcomes for peritonitis. Improvement in outcome will be determined by scores such as MOF, SOFA and survival.
2. Identification of biomarkers (including immunoglobulin levels, HLA-DR, NF-kB1 and other immunological biomarkers) to identify patient subpopulations that benefit most from IgGAM treatment. These patients will form the basis for a further randomized, controlled, double-blind Phase III trial (RCT) to demonstrate the benefit of this treatment.
3. In addition, these biomarkers could help to guide a targeted, i.e. "personalized", adjuvant therapy with Pentaglobin® (IgGAM) in the indication of peritonitis.

DETAILED DESCRIPTION:
The aim of this prospective, randomized, controlled trial is to provide evidence for adjuvant IgGAM treatment with regard to

1. Improvement of patient outcomes for peritonitis. Improvement in outcome will be determined by scores such as MOF, SOFA and survival.
2. Identification of biomarkers (including immunoglobulin levels, HLA-DR, NF-kB1 and other immunological biomarkers) to identify patient subpopulations that benefit most from IgGAM treatment. These patients will form the basis for a further randomized, controlled, double-blind Phase III trial (RCT) to demonstrate the benefit of this treatment.
3. In addition, these biomarkers could help to guide a targeted, i.e. "personalized", adjuvant therapy with Pentaglobin® (IgGAM) in the indication of peritonitis.

The control group receives Standard-of-Care treatment. The intervention group is additionally treated with IgGAM (Pentaglobin®) as an add-on treatment to Standard-of-Care.

Pentaglobin® is administered by continuous intravenous infusion over a period of 5 days of 0.4 ml/kg body weight/hour until the total dose of 7 ml/kg body weight/day is reached.

Primary outcome: Change in Multiple Organ Failure (MOF) score (measured in lung, heart, kidney, liver, blood) from baseline to day 7 after surgical infectious source control in the context of peritonitis.

The MOF score is determined in the morning. The following score points are distributed per organ: Normal organ function: 0 score points; organ dysfunction: 1 score point; single organ failure: 2 score points. A score > 4 in the sum of the 5 organs indicates multiple organ failure. Patients who died before the MOF score was obtained are assigned a score of 10 score points.

Secondary outcome:

* Death within 28 days
* Death within 90 days
* Change in MOF score from baseline to day 5
* Multi-Organ Failure ( > 4 MOF score points on day 7)

Exploratory objectives:

* Effects of Pentaglobin® therapy on the SOFA score (determined in the organs lung, CNS, circulation, liver, coagulation and kidney).
* Interaction of the biomarkers "NF-kB1" (steady), "CRP (≥ 70 mg/L), IgA (< 150 mg/dl), IgG (< 700 mg/dl), IgM (< 35 mg/dl) and HLA-DR expression (≤ 8,000 molecules per monocyte) with therapy in terms of change in MOF score from baseline to days 5 and 7 and death within 28 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is diagnosed with secondary or quaternary peritonitis
2. The time of the surgical infectious source control is within 6 hours of indication (defined as date and time of registration for surgical or minimal invasive procedure).
3. Sepsis and / or septic shock (according to the current sepsis guideline of the German Sepsis Society).
4. SOFA Score ≥ 8
5. The concentration of IL-6 is ≥ 1000 pg / ml
6. Treatment with antibiotics is started within 12 hours of admission to the Intensive Care Unit
7. The informed consent form has been signed by the patient and / or by his legal representative (such as his spouse, an health care proxy authorized or a legal representative) or by a consultant physician

Exclusion criteria

1. Patients with a life expectancy of less than 90 days due to medical conditions unrelated to peritonitis nor with sepsis and / or septic shock.
2. For female patients: The patient is pregnant or breastfeeding.
3. The patient is a minor (< 18 years of age).
4. The patient has known chronic renal dysfunction requiring dialysis (creatinine ≥ 3.4 mg / dl or creatinine clearance ≤ 30 mL/min/1.73 m²).
5. The patient has acute, primarily non-infectious pancreatitis or mediastinitis.
6. The patient has a BMI > 40.
7. The patient has any contraindication to study drug.
8. The patient has participated in another clinical trial within the last 30 days.
9. The patient is in a dependent or employment relationship with the sponsor or investigator.
10. The patient is institutionalized by court or government order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in Multiple Organ Failure (MOF) score (measured in lung, heart, kidney, liver, blood) from baseline to day 7 after surgical infectious source control in the context of peritonitis. | 7 days
  The MOF score is determined in the morning. The following points are distributed per organ: Normal organ function: 0 points; organ dysfunction: 1 point; single organ failure: 2 points. A score > 4 in the sum of the 5 organs indicates multiple organ failure. Patients who died before the MOF score are assigned a score of 10 points.

SECONDARY OUTCOMES:
Death within 28 days | 28 days
  Evaluation of death within 28-days.
Death within 90 days | 90 days
  Evaluation of death within 90-days.
Change in MOF Score from baseline to day 5 | 5 days
  Change in MOF Score from baseline to day 5.
Multi-Organ Failure (i.e., > 4 MOF points) on day 7 | 7 days
  MOF (i.e., > 4 MOF points) on day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Marx, Univ.-Prof., Principal Investigator — RWTH Aachen University
Locations (20):
- Medizinische Universität Wien, Klinische Abteilung für Allgemeine Anästhesie und Intensivmedizin, Vienna, Austria
- Germany (19):
  - Universitätsklinikum Tübingen, Universitätsklinik für Anästhesiologie und Intensivmedizin, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Regensburg, Klinik für Anästhesiologie, Regensburg, Bavaria
  - Universitätsklinikum Essen, Klinik für Anästhesiologie und Intensivmedizin, Essen, North Rhine-Westphalia
  - Charité - Universitätsmedizin Berlin, Klinik für Anästhesiologie mit Schwerpunkt operative Intensivmedizin, Berlin, State of Berlin
  - Uniklinik RWTH Aachen, Klinik für Operative Intensivmedizin und Intermediate Care, Aachen
  - Universitätsklinikum Knappschaftskrankenhaus Bochum GmbH, Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie, Bochum
  - Klinikum Westfalen, Knappschaftskrankenhaus Dortmund, Klinik für Anästhesiologie, operative Intensivmedizin und Schmerztherapie, Dortmund
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Anästhesiologie und Intensivtherapie, Dresden
  - Universitätsklinikum Düsseldorf, Klinik für Anästhesiologie, Düsseldorf
  - Universitätklinikum Frankfurt, Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie, Frankfurt
  - Universitätsklinikum Freiburg, Klinik für Allgemein- und Viszeralchirurgie, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Intensivmedizin, Hamburg
  - Medizinische Hochschule Hannover, Zentrum für Anästhesiologie und Intensivmedizin, Hanover
  - Universitätsklinikum Heidelberg, Anästhesiologische Klinik, Heidelberg
  - Klinikum Magdeburg, Klinik für Intensivmedizin, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, Mainz
  - Klinikum der Universität München, Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, München
  - Klinikum Nürnberg, Klinik für Anästhesiologie und operative Intensivmedizin, Nuremberg
  - Heinrich-Braun-Klinikum gGmbH, Klinik für Anästhesie, Intensivmedizin, Notfallmedizin und Schmerztherapie, Zwickau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kujath P., Rodloff Peritonitis UNI-MED, 2001 ISBN 3-8999-549-5
- [Background] Chang HJ, Lynm C, Glass RM. JAMA patient page. Sepsis. JAMA. 2010 Oct 27;304(16):1856. doi: 10.1001/jama.304.16.1856. No abstract available. PMID 20978264
- [Background] Harbarth S, Holeckova K, Froidevaux C, Pittet D, Ricou B, Grau GE, Vadas L, Pugin J; Geneva Sepsis Network. Diagnostic value of procalcitonin, interleukin-6, and interleukin-8 in critically ill patients admitted with suspected sepsis. Am J Respir Crit Care Med. 2001 Aug 1;164(3):396-402. doi: 10.1164/ajrccm.164.3.2009052. PMID 11500339
- [Background] Heyland DK, Muscedere J, Drover J, Jiang X, Day AG; Canadian Critical Care Trials Group. Persistent organ dysfunction plus death: a novel, composite outcome measure for critical care trials. Crit Care. 2011;15(2):R98. doi: 10.1186/cc10110. Epub 2011 Mar 18. PMID 21418560
- [Background] Muller B, Becker KL, Schachinger H, Rickenbacher PR, Huber PR, Zimmerli W, Ritz R. Calcitonin precursors are reliable markers of sepsis in a medical intensive care unit. Crit Care Med. 2000 Apr;28(4):977-83. doi: 10.1097/00003246-200004000-00011. PMID 10809269
- [Background] Maruna P, Nedelnikova K, Gurlich R. Physiology and genetics of procalcitonin. Physiol Res. 2000;49 Suppl 1:S57-61. PMID 10984072
- [Background] Clec'h C, Fosse JP, Karoubi P, Vincent F, Chouahi I, Hamza L, Cupa M, Cohen Y. Differential diagnostic value of procalcitonin in surgical and medical patients with septic shock. Crit Care Med. 2006 Jan;34(1):102-7. doi: 10.1097/01.ccm.0000195012.54682.f3. PMID 16374163
- [Background] Monneret G, Doche C, Durand DV, Lepape A, Bienvenu J. Procalcitonin as a specific marker of bacterial infection in adults. Clin Chem Lab Med. 1998 Jan;36(1):67-8. doi: 10.1515/CCLM.1998.012. No abstract available. PMID 9594089
- [Background] Brunkhorst FM. [Sepsismarker--what is useful?]. Dtsch Med Wochenschr. 2008 Nov;133(48):2512-5. doi: 10.1055/s-0028-1100949. Epub 2008 Nov 19. No abstract available. German. PMID 19021084
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Background] Van Snick J. Interleukin-6: an overview. Annu Rev Immunol. 1990;8:253-78. doi: 10.1146/annurev.iy.08.040190.001345. No abstract available. PMID 2188664
- [Background] Panacek EA, Marshall JC, Albertson TE, Johnson DH, Johnson S, MacArthur RD, Miller M, Barchuk WT, Fischkoff S, Kaul M, Teoh L, Van Meter L, Daum L, Lemeshow S, Hicklin G, Doig C; Monoclonal Anti-TNF: a Randomized Controlled Sepsis Study Investigators. Efficacy and safety of the monoclonal anti-tumor necrosis factor antibody F(ab')2 fragment afelimomab in patients with severe sepsis and elevated interleukin-6 levels. Crit Care Med. 2004 Nov;32(11):2173-82. doi: 10.1097/01.ccm.0000145229.59014.6c. PMID 15640628
- [Background] Kuster H, Weiss M, Willeitner AE, Detlefsen S, Jeremias I, Zbojan J, Geiger R, Lipowsky G, Simbruner G. Interleukin-1 receptor antagonist and interleukin-6 for early diagnosis of neonatal sepsis 2 days before clinical manifestation. Lancet. 1998 Oct 17;352(9136):1271-7. doi: 10.1016/S0140-6736(98)08148-3. PMID 9788457
- [Background] Meisel C, Schefold JC, Pschowski R, Baumann T, Hetzger K, Gregor J, Weber-Carstens S, Hasper D, Keh D, Zuckermann H, Reinke P, Volk HD. Granulocyte-macrophage colony-stimulating factor to reverse sepsis-associated immunosuppression: a double-blind, randomized, placebo-controlled multicenter trial. Am J Respir Crit Care Med. 2009 Oct 1;180(7):640-8. doi: 10.1164/rccm.200903-0363OC. Epub 2009 Jul 9. PMID 19590022
- [Background] Schefold JC, von Haehling S, Corsepius M, Pohle C, Kruschke P, Zuckermann H, Volk HD, Reinke P. A novel selective extracorporeal intervention in sepsis: immunoadsorption of endotoxin, interleukin 6, and complement-activating product 5a. Shock. 2007 Oct;28(4):418-25. doi: 10.1097/shk.0b013e31804f5921. PMID 17558345
- [Background] Bermejo-Martin JF, Rodriguez-Fernandez A, Herran-Monge R, Andaluz-Ojeda D, Muriel-Bombin A, Merino P, Garcia-Garcia MM, Citores R, Gandia F, Almansa R, Blanco J; GRECIA Group (Grupo de Estudios y Analisis en Cuidados Intensivos). Immunoglobulins IgG1, IgM and IgA: a synergistic team influencing survival in sepsis. J Intern Med. 2014 Oct;276(4):404-12. doi: 10.1111/joim.12265. Epub 2014 May 29. PMID 24815605
- [Background] Giamarellos-Bourboulis EJ, Apostolidou E, Lada M, Perdios I, Gatselis NK, Tsangaris I, Georgitsi M, Bristianou M, Kanni T, Sereti K, Kyprianou MA, Kotanidou A, Armaganidis A; Hellenic Sepsis Study Group. Kinetics of circulating immunoglobulin M in sepsis: relationship with final outcome. Crit Care. 2013 Oct 21;17(5):R247. doi: 10.1186/cc13073. PMID 24144038
- [Background] Tamayo E, Fernandez A, Almansa R, Carrasco E, Goncalves L, Heredia M, Andaluz-Ojeda D, March G, Rico L, Gomez-Herreras JI, de Lejarazu RO, Bermejo-Martin JF. Beneficial role of endogenous immunoglobulin subclasses and isotypes in septic shock. J Crit Care. 2012 Dec;27(6):616-22. doi: 10.1016/j.jcrc.2012.08.004. Epub 2012 Oct 22. PMID 23089676
- [Background] Koo DJ, Zhou M, Chaudry IH, Wang P. The role of adrenomedullin in producing differential hemodynamic responses during sepsis. J Surg Res. 2001 Feb;95(2):207-18. doi: 10.1006/jsre.2000.6013. PMID 11162047
- [Background] Wang P, Ba ZF, Cioffi WG, Bland KI, Chaudry IH. The pivotal role of adrenomedullin in producing hyperdynamic circulation during the early stage of sepsis. Arch Surg. 1998 Dec;133(12):1298-304. doi: 10.1001/archsurg.133.12.1298. PMID 9865646
- [Background] Marino R, Struck J, Maisel AS, Magrini L, Bergmann A, Di Somma S. Plasma adrenomedullin is associated with short-term mortality and vasopressor requirement in patients admitted with sepsis. Crit Care. 2014 Feb 17;18(1):R34. doi: 10.1186/cc13731. PMID 24533868
- [Background] Ueda S, Nishio K, Minamino N, Kubo A, Akai Y, Kangawa K, Matsuo H, Fujimura Y, Yoshioka A, Masui K, Doi N, Murao Y, Miyamoto S. Increased plasma levels of adrenomedullin in patients with systemic inflammatory response syndrome. Am J Respir Crit Care Med. 1999 Jul;160(1):132-6. doi: 10.1164/ajrccm.160.1.9810006. PMID 10390390
- [Background] Adamzik M, Frey UH, Mohlenkamp S, Scherag A, Waydhas C, Marggraf G, Dammann M, Steinmann J, Siffert W, Peters J. Aquaporin 5 gene promoter--1364A/C polymorphism associated with 30-day survival in severe sepsis. Anesthesiology. 2011 Apr;114(4):912-7. doi: 10.1097/ALN.0b013e31820ca911. PMID 21427539
- [Background] Zhu Y, Qiu HB, Liu JT, Wang Y, Lin HY, Xu Y, Jiang L, Shi Y, Zhu X, Ning B, Cheng R, Xie ZY, Ma PL. [Effect of endothelial nitric oxide synthase gene polymorphisms upon disease severity and outcome in septic patients]. Zhonghua Yi Xue Za Zhi. 2010 Apr 6;90(13):906-11. Chinese. PMID 20646511
- [Background] Thair SA, Walley KR, Nakada TA, McConechy MK, Boyd JH, Wellman H, Russell JA. A single nucleotide polymorphism in NF-kappaB inducing kinase is associated with mortality in septic shock. J Immunol. 2011 Feb 15;186(4):2321-8. doi: 10.4049/jimmunol.1002864. Epub 2011 Jan 21. PMID 21257964
- [Background] Beyer K, Menges P, Kessler W, Heidecke CD. [Pathophysiology of peritonitis]. Chirurg. 2016 Jan;87(1):5-12. doi: 10.1007/s00104-015-0117-6. German. PMID 26661744
- [Background] Rodriguez A, Rello J, Neira J, Maskin B, Ceraso D, Vasta L, Palizas F. Effects of high-dose of intravenous immunoglobulin and antibiotics on survival for severe sepsis undergoing surgery. Shock. 2005 Apr;23(4):298-304. doi: 10.1097/01.shk.0000157302.69125.f8. PMID 15803051
- [Background] Cavazzuti I, Serafini G, Busani S, Rinaldi L, Biagioni E, Buoncristiano M, Girardis M. Early therapy with IgM-enriched polyclonal immunoglobulin in patients with septic shock. Intensive Care Med. 2014 Dec;40(12):1888-96. doi: 10.1007/s00134-014-3474-6. Epub 2014 Sep 13. PMID 25217146
- [Background] Alejandria MM, Lansang MA, Dans LF, Mantaring JB 3rd. Intravenous immunoglobulin for treating sepsis, severe sepsis and septic shock. Cochrane Database Syst Rev. 2013 Sep 16;2013(9):CD001090. doi: 10.1002/14651858.CD001090.pub2. PMID 24043371
- [Background] Janssens U. [Treatment of sepsis and septic shock with immunoglobulins]. Dtsch Med Wochenschr. 2014 Jan;139(5):178. doi: 10.1055/s-0032-1329177. Epub 2014 Jan 21. No abstract available. German. PMID 24449349
- [Background] Reinhart K, Brunkhorst FM, Bone HG, Bardutzky J, Dempfle CE, Forst H, Gastmeier P, Gerlach H, Grundling M, John S, Kern W, Kreymann G, Kruger W, Kujath P, Marggraf G, Martin J, Mayer K, Meier-Hellmann A, Oppert M, Putensen C, Quintel M, Ragaller M, Rossaint R, Seifert H, Spies C, Stuber F, Weiler N, Weimann A, Werdan K, Welte T; German Interdisciplinary Association for Intensive and Emergency Care Medicine; German Sepsis Society. [Prevention, diagnosis, treatment, and follow-up care of sepsis. First revision of the S2k Guidelines of the German Sepsis Society (DSG) and the German Interdisciplinary Association for Intensive and Emergency Care Medicine (DIVI)]. Anaesthesist. 2010 Apr;59(4):347-70. doi: 10.1007/s00101-010-1719-5. No abstract available. German. PMID 20414762
- [Background] Goris RJ, te Boekhorst TP, Nuytinck JK, Gimbrere JS. Multiple-organ failure. Generalized autodestructive inflammation? Arch Surg. 1985 Oct;120(10):1109-15. doi: 10.1001/archsurg.1985.01390340007001. PMID 4038052
- [Background] Lefering R, Goris RJ, van Nieuwenhoven EJ, Neugebauer E. Revision of the multiple organ failure score. Langenbecks Arch Surg. 2002 Apr;387(1):14-20. doi: 10.1007/s00423-001-0269-3. Epub 2002 Jan 31. PMID 11981679
- [Background] Casserly B, Phillips GS, Schorr C, Dellinger RP, Townsend SR, Osborn TM, Reinhart K, Selvakumar N, Levy MM. Lactate measurements in sepsis-induced tissue hypoperfusion: results from the Surviving Sepsis Campaign database. Crit Care Med. 2015 Mar;43(3):567-73. doi: 10.1097/CCM.0000000000000742. PMID 25479113
- [Background] Weigelt JA. Empiric treatment options in the management of complicated intra-abdominal infections. Cleve Clin J Med. 2007 Aug;74 Suppl 4:S29-37. doi: 10.3949/ccjm.74.suppl_4.s29. PMID 17847176
- [Background] Wong PF, Gilliam AD, Kumar S, Shenfine J, O'Dair GN, Leaper DJ. Antibiotic regimens for secondary peritonitis of gastrointestinal origin in adults. Cochrane Database Syst Rev. 2005 Apr 18;2005(2):CD004539. doi: 10.1002/14651858.CD004539.pub2. PMID 15846719
- [Background] Mebazaa A, Laterre PF, Russell JA, Bergmann A, Gattinoni L, Gayat E, Harhay MO, Hartmann O, Hein F, Kjolbye AL, Legrand M, Lewis RJ, Marshall JC, Marx G, Radermacher P, Schroedter M, Scigalla P, Stough WG, Struck J, Van den Berghe G, Yilmaz MB, Angus DC. Designing phase 3 sepsis trials: application of learned experiences from critical care trials in acute heart failure. J Intensive Care. 2016 Mar 31;4:24. doi: 10.1186/s40560-016-0151-6. eCollection 2016. PMID 27034779
- [Derived] Kalvelage C, Zacharowski K, Bauhofer A, Gockel U, Adamzik M, Nierhaus A, Kujath P, Eckmann C, Pletz MW, Bracht H, Simon TP, Winkler M, Kindgen-Milles D, Albertsmeier M, Weigand M, Ellger B, Ragaller M, Ullrich R, Marx G. Personalized medicine with IgGAM compared with standard of care for treatment of peritonitis after infectious source control (the PEPPER trial): study protocol for a randomized controlled trial. Trials. 2019 Mar 4;20(1):156. doi: 10.1186/s13063-019-3244-4. PMID 30832742